CLINICAL TRIAL: NCT01286116
Title: A MULTINATIONAL TRIAL TO EVALUATE THE PARACHUTE IMPLANT SYSTEM: PARACHUTE PercutAneous Ventricular RestorAtion in Chronic Heart FailUre Due to Ischemic HearT DiseasE
Brief Title: A Multinational Trial To Evaluate The Parachute Implant System
Acronym: PARACHUTE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company closed
Sponsor: CardioKinetix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA0444
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: heart failure; percutaneous; interventional cardiology; apical remodeling; LV dilatation; akinesis; dyskinesis; myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Parachute implant
  Interventions: Device: Parachute Implant

INTERVENTIONS:
Device: Parachute Implant — Mechanical ventricular partitioning

SUMMARY:
The primary objective is to assess the safety of the CardioKinetix Parachute Implant and Delivery System in the partitioning of the left ventricle in patients with heart failure due to ischemic heart disease.

DETAILED DESCRIPTION:
While current therapies for heart failure (including but not limited to: medical management, cardiac resynchronization and ICDs) may represent the best treatment available today for the majority of HF patients, the medical community recognizes that pharmacologic therapy has been optimized to nearly the extent that is possible, and that any incremental improvements in the management of HF patients will now come from device based therapies. With this background, CardioKinetix has developed a catheter-based intravascular approach to ventricular partitioning using an implantable device. The purpose of this study is to assess the safety of using the CardioKinetix Parachute device to isolate the malfunctioning portion of the left ventricle in patients with symptoms of HF due to ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study must meet ALL of the following inclusion criteria:

  1. Akinesis or dyskinesis due to myocardial infarction limited to anteroapical region
  2. Subject is not hospitalized at time of enrollment.
  3. Diagnosis of heart failure for a minimum of 6 months prior to enrollment
  4. NYHA Class at time of enrollment, either:

     * NYHA Class III or Ambulatory IV - if predominant during the 3-month period prior to enrollment
     * NYHA Class II - if diagnosed with NYHA Class III or IV during 3-month period prior to enrollment
  5. LVEF >15% and ≤ 40% as measured by echocardiography.
  6. Post LV MI structural heart dysfunction represented by LV wall motion abnormality (WMA) by echocardiography.
  7. Eligible for cardiac surgery
  8. Between 18 and 79 years of age (inclusive)
  9. Receiving appropriate medical treatment for heart failure according to the ACC/AHA 2009 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult during the three months prior to enrollment
  10. Female patients with childbearing potential must have a negative pregnancy test (within 7 days of the procedure) and must agree not to attempt to become pregnant during the course of the study
  11. Provide written informed consent
  12. Agree to the protocol-required follow-up

Exclusion Criteria:

Candidates will be excluded from the study if ANY of the following conditions apply:

1. Untreated clinically significant coronary artery disease requiring intervention.
2. Acute MI (see MI definition) within 60 days of enrollment or patients with suspected evolving MI at time of enrollment
3. Cardiogenic shock within 72 hours of enrollment
4. Revascularization procedure (PCI or CABG) within 60 days of enrollment
5. Patient has received a pacemaker, ICD, or CRT device within 60 days of enrollment
6. Moderate aortic stenosis and regurgitation (aortic or mitral) >2+.
7. History of aborted sudden cardiac death, if patient has not received an ICD and has potentially lethal ventricular arrhythmia, VT or VF
8. A known hypersensitivity or contraindication to aspirin, heparin, warfarin, nitinol (titanium and nickel alloy), or sensitivity to contrast media, which cannot be adequately pre medicated.
9. Aortic valve replacement or repair
10. Blood dyscrasia, history of bleeding diathesis or coagulopathy, or hypercoagulable states.
11. Active peptic ulcer or GI bleeding within the past 3 months
12. Patient has suffered a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
13. History of Kawasaki's disease
14. Patient has received a heart, lung, liver and/or kidney transplant
15. Patient on dialysis or expected to require hemodialysis within 12 months
16. Patient has chronic liver disease
17. Impaired renal function that places patient at risk of contrast induced renal failure
18. Ongoing sepsis, including active endocarditis.
19. Co-morbidities associated with a life expectancy of less than 12-months or there are factors making echo and clinical follow-up difficult (no permanent address, etc.)
20. Patient is currently participating in another investigational device or drug research study for which the follow-up period is not complete

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The successful delivery and deployment of the Parachute Implant through 6-month follow-up without the occurrence of Major Adverse Cardiac Events (MACE) | 6-months
  Assessment of safety defined as the successful delivery and deployment of the Parachute Implant through 6-month follow-up without the occurrence of Major Adverse Cardiac Events (MACE) related to the investigational device.

SECONDARY OUTCOMES:
Change in Left Ventricular Volume Indexes. | 6 months
  Change in Left Ventricular Volume Indexes including End Systolic {LVESVI} and End Diastolic {LVEDVI}) measured by echocardiography from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Thomas, MD, Principal Investigator — St. Thomas' Hospital
Locations (13):
- France (2):
  - Hospital of Cardiology Louis Pradel (Lyon), Bron
  - Institut Cardiovasculaire Paris-Sud, Massy
- Germany (2):
  - University of Heidelberg, Heidelberg
  - Universitat Rostock, Rostock
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- University of Amsterdam AMC, Amsterdam, Netherlands
- Portugal (2):
  - Hospital Santa Marta, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Clinical Center of Serbia (KCS), Belgrade, Serbia
- Ljubljana University Medical Center (Univerzitetni Klinicni Center Ljubljana), Ljubljana, Slovenia
- United Kingdom (3):
  - Papworth Hospital, Cambridge
  - St. Thomas' Hospital, London
  - University College of London (The Heart Hospital), London

REFERENCES:
- [Derived] Costa MA, Mazzaferri EL Jr, Sievert H, Abraham WT. Percutaneous ventricular restoration using the parachute device in patients with ischemic heart failure: three-year outcomes of the PARACHUTE first-in-human study. Circ Heart Fail. 2014 Sep;7(5):752-8. doi: 10.1161/CIRCHEARTFAILURE.114.001127. Epub 2014 Jul 18. PMID 25037310
- [Derived] Costa MA, Pencina M, Nikolic S, Engels T, Templin B, Abraham WT. The PARACHUTE IV trial design and rationale: percutaneous ventricular restoration using the parachute device in patients with ischemic heart failure and dilated left ventricles. Am Heart J. 2013 Apr;165(4):531-6. doi: 10.1016/j.ahj.2012.12.022. Epub 2013 Feb 19. PMID 23537969